CLINICAL TRIAL: NCT04155411
Title: Efficacy and Safety of Dasatinib 70 mg as First-Line Treatment for Newly Diagnosed Chronic-Phase Chronic Myeloid Leukemia (CML-CP)
Brief Title: Dose Reduced Dasatinib (70 mg Daily) as First-line Treatment for Newly Diagnosed CML-CP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20191103
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-06

CONDITIONS: Dasatinib; BCR-ABL; Chronic Myeloid Leukemia
Keywords: Dasatinib, CML-CP
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dasatinib 70 mg (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 70 mg of Dasatinib orally daily for 12 months

SUMMARY:
The purpose of this study is to explore the efficacy and safety of dasatinib 70 mg once daily as first line therapy in patients with early chronic phase (CP) chronic myeloid leukemia (CML).

DETAILED DESCRIPTION:
A multicenter, single-arm, prospective, open-label study to detect the efficacy and safety of 70mg dasatinib by measuring rates of major molecular response (MMR) at 12 months in patients with CML-CP in China. Approximately 65 Patients will be recruited consecutively from the study sites during the enrollment period and will be given dasatinib 70 mg QD. The duration of patient participation will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of Ph+ or BCR-ABL positive CML-CP within 6 months.
* ECOG performance of 0-2.
* Adequate end organ function defined as the following: total bilirubin <1.5x ULN, SGPT <2.5x ULN, creatinine <1.5x ULN.
* Patients must sign an informed consent form (ICF) indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital

Exclusion Criteria:

* History of any TKI treatments.
* History of Pulmonary arterial hypertension and Pleural effusion
* NYHA cardiac class 3-4 heart disease.
* Cardiac symptoms - Patients meeting the following criteria are not eligible unless cleared by a cardiologist:
* Uncontrolled angina within 12 months.
* Diagnosed or suspected congenital long QT syndrome.
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes).
* Prolonged QTc interval on pre-entry electrocardiogram (>450 msec).
* Patients with active uncontrolled psychiatric disorders including: psychosis, major depression, and bipolar disorders.
* Women of pregnancy potential must practice an effective method of birth control, unless otherwise instructed, during the course of the study in a manner such that risk of failure is minimized.
* Pregnant or breast-feeding women are excluded.
* Patients in late chronic phase (i.e. time from diagnosis to treatment >12 months), accelerated phase (except as noted in inclusion criteria 2) or blast phase are excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve and maintain MMR at 12 months using RQ-PCR test | 12 months
  Major molecular response (MMR) is defined as BCR-ABL1 ≤ 0.1%

SECONDARY OUTCOMES:
Proportion of patients with MR 4.0 at 12 months. | 12 months
  Molecular response (MR) 4.0 is defined as BCR-ABL transcripts ≤ 0.01%
Proportion of patients with MR 4.5 at 12 months. | 12 months
  Molecular response (MR) 4.5 is defined as BCR-ABL transcripts ≤ 0.0032%
Proportion of patients with Complete cytogenetic response (CCyR) at 12 months | 12 months
  defined as 0% Ph+ metaphases, or FISH ≤2%, or BCR-ABL transcripts (IS) ≤1%
Incidence of adverse events (AEs) and serious adverse events (SAEs) to dasatinib | 18 months
  Evaluation of adverse events (AEs), serious AEs (SAEs), and clinically relevant changes in laboratory tests according to laboratory reference ranges

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Du, Shenzhen, Guangdong, China